CLINICAL TRIAL: NCT05275270
Title: Role of Topical Oxytocin Gel On Vaginal Atrophy, Psycho-sexual and Psychological Function and Metabolic and Inflammatory Parameters in Post-Menopausal Egyptian Women
Brief Title: Role of Topical Oxytocin Gel in Post-Menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Collaborators: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Asem Anwar Moussa, Professor, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Topical Oxytocin Gel
Record Dates: First submitted 2022-02-22; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Menopause Related Conditions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): patients were treated with an active gel containing oxytocin
  Interventions: Other: oxytocin gel
- Group B (Placebo Comparator): patients were treated with placebo gel without oxytocin
  Interventions: Other: placebo gel

INTERVENTIONS:
Other: oxytocin gel — The active oxytocin gel (A) consisted of oxytocin dissolved in a gel-based on hypromellose with a pH of 3.8. 1 ml of gel contained 600 IU of oxytocin
  Arms: Group A
Other: placebo gel — The placebo gel (B) consisted of the gel alone
  Arms: Group B

SUMMARY:
Aim of the current study:

To evaluate the effect of a14 day treatment period with local intravaginal application of an oxytocin-containing gel on vaginal atrophy, psychosexual and psychological/cognitive function, and metabolic, stress, and inflammatory parameters in Egyptian post-menopausal women

ELIGIBILITY:
Inclusion Criteria:

* The women were post-menopausal and were between 47 and 67 years old
* The women's last menstruation had occurred more than one year prior to the study
* The women had an established vaginal atrophy
* The women scored < 26 in the Female Sexual Function Index (FSFI)
* The women had an active sexual relationship

Exclusion Criteria:

* Women who smoked
* Women who used hormone replacement therapy
* Women using a vaginal lubricant
* Women having any vaginal bleeding or any breast diseases
* Women having any undiagnosed genitalia disorder
* Women suffering from chronic diseases such as diabetes, hypertension, cardiovascular disease, or psychiatric disease

Ages: 47 Years to 66 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
vaginal pallor | by the end of 14 successive days of regular use
  A vaginal inspection was performed to establish the presence of vaginal pallor
intravaginal potential of hydrogen (pH) | by the end of 14 successive days of regular use
  Intravaginal pH was measured by a litmus paper applied intravaginally
Cytological examination of vaginal smear | by the end of 14 successive days of regular use
  A piece of cotton was applied on a stick ( a vaginal swab) to the posterior vaginal wall to collect material from the epithelium
The Female Sexual Function Index (FSFI) questionnaire | by the end of 14 successive days of regular use
  19 questions to measure sexual function in six domains, including sexual desire, arousal, lubrication, orgasm, satisfaction, and pain. We applied the modified FSFI, which included 6 questions to measure sexual function in the six domains (one question for each). The score for each domain is evaluated by six levels (from 0 to 6); the lowest is 0, and the maximum is 6. The sexual function was assessed by the sum of all 6 domains.
questionnaire to assess the psychological function | by the end of 14 successive days of regular use
  It consisted of 6 domains, including social cognition, memory, social trust, prosocial behavior, aggressive behavior, and depression, which included 2 questions for memory and depression and one question for social cognition, social trust, prosocial behavior, and aggressive behavior. The score for each domain is evaluated by 4 levels (from 0 to 3), the lowest is 0, and the maximum is 3. The psychological function was assessed by the sum of all domains.
Visual Analogue Scale (VAS) | by the end of 14 successive days of regular use
  to assess the severity of the vaginal pain if present. The score ranges from 0 if no pain to 10 for the severest degree of pain.
Cholesterol | by the end of 14 successive days of regular use
  to assess the serum level in both groups
Triglyceride | by the end of 14 successive days of regular use
  to assess the serum level in both groups
HDL-C | by the end of 14 successive days of regular use
  to assess the serum level in both groups
LDL-C | by the end of 14 successive days of regular use
  to assess the serum level in both groups
C-Reactive Protein (CRP) | by the end of 14 successive days of regular use
  to assess the serum level in both groups
Random blood sugar (RBS) | by the end of 14 successive days of regular use
  to assess the serum level in both groups
HBA1C | by the end of 14 successive days of regular use
  to assess the serum level in both groups
Insulin | by the end of 14 successive days of regular use
  to assess the serum level in both groups
C-Peptide F | by the end of 14 successive days of regular use
  to assess the serum level in both groups
Cortisol at morning | by the end of 14 successive days of regular use
  to assess the serum level in both groups
Interleukin-6 (IL-6) | by the end of 14 successive days of regular use
  to assess the serum level in both groups
Tumor necrosis factor-Alfa (TNF-Alfa) | by the end of 14 successive days of regular use
  to assess the serum level in both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Galaa Teaching Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moussa A, Moberg KU, Elgrahy I, Elsayied M, Abdel-Rasheed M, Farouk M, Saad H, Meshaal H. Effect of topical oxytocin gel on vaginal mucosa in postmenopausal Egyptian women: a clinical randomized trial. J Sex Med. 2023 Feb 14;20(2):177-183. doi: 10.1093/jsxmed/qdac021. PMID 36763919